CLINICAL TRIAL: NCT00572455
Title: A 2-STAGE, PHASE 2, DOUBLE-MASKED, RANDOMIZED, VEHICLE CONTROLLED, DOSE RESPONSE TRIAL OF PF-04217329 AND THE MARKETED FORMULATION OF LATANOPROST IN PATIENTS WITH PRIMARY OPEN ANGLE GLAUCOMA OR OCULAR HYPERTENSION
Brief Title: Safety and Efficacy of PF-04217329 in Patients With Glaucoma or Elevated Eye Pressure.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0191001
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Primary Open-Angle Glaucoma; Ocular Hypertension
Keywords: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — PF 04217329; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (14):
- Stage 1: PF-04217329 - Lowest Dose (Experimental)
  Interventions: Drug: PF-04217329 - Lowest Dose
- Stage 1: PF-04217329 - Low Dose (Experimental)
  Interventions: Drug: PF-04217329 - Low Dose
- Stage 1: PF-04217329 - Middle Dose (Experimental)
  Interventions: Drug: PF-04217329 - Middle Dose
- Stage 1: PF-04217329 - High Middle Dose (Experimental)
  Interventions: Drug: PF-04217329 - High Middle Dose
- Stage 1: PF-04217329 - High Dose (Experimental)
  Interventions: Drug: PF-04217329 - High Dose
- Stage 1: PF-02417329 - Highest Dose (Experimental)
  Interventions: Drug: PF-4217329 - Highest Dose
- Stage 1: PF-04217329 - Vehicle (Experimental)
  Interventions: Drug: PF-04217329 - Vehicle
- Stage 2: PF-04217329 - Low Dose + Latanoprost Vehicle (Experimental)
  Interventions: Drug: Latanoprost Vehicle; Drug: PF-04217329 - Low Dose
- Stage 2: PF-04217329 - Middle Dose + Latanoprost Vehicle (Experimental)
  Interventions: Drug: Latanoprost Vehicle; Drug: PF-04217329 - Middle Dose
- Stage 2: PF-04217329 - High Dose + Latanoprost Vehicle (Experimental)
  Interventions: Drug: Latanoprost Vehicle; Drug: PF-04217329 - High Dose
- Stage 2: PF-04217329 - Low Dose + Latanoprost 0.005% (Experimental)
  Interventions: Drug: Latanoprost 0.005%; Drug: PF-04217329 - Low Dose
- Stage 2: PF-04217329 - Middle Dose + Latanoprost 0.005% (Experimental)
  Interventions: Drug: Latanoprost 0.005%; Drug: PF-04217329 - Middle Dose
- Stage 2: PF-04217329 - High Dose + Latanoprost 0.005% (Experimental)
  Interventions: Drug: Latanoprost 0.005%; Drug: PF-04217329 - High Dose
- Stage 2: PF-04217329 - Vehicle + Latanoprost 0.005% (Experimental)
  Interventions: Drug: Latanoprost 0.005%; Drug: PF-04217329 - Vehicle

INTERVENTIONS:
Drug: PF-04217329 - Lowest Dose — 1 drop of lowest dose PF-04217329, once a day, per dosed eye for duration of study.
  Arms: Stage 1: PF-04217329 - Lowest Dose
Drug: PF-04217329 - Low Dose — 1 drop of low dose PF-04217329, once a day, per dosed eye for duration of study.
  Arms: Stage 1: PF-04217329 - Low Dose
Drug: PF-04217329 - Middle Dose — 1 drop of middle dose PF-04217329, once a day, per dosed eye for duration of study.
  Arms: Stage 1: PF-04217329 - Middle Dose
Drug: PF-04217329 - High Middle Dose — 1 drop of high middle dose PF-04217329, once a day, per dosed eye for duration of study.
  Arms: Stage 1: PF-04217329 - High Middle Dose
Drug: PF-04217329 - High Dose — 1 drop of high dose PF-04217329, once a day, per dosed eye for duration of study.
  Arms: Stage 1: PF-04217329 - High Dose
Drug: PF-4217329 - Highest Dose — 1 drop of highest dose PF-04217329, once a day, per dosed eye for duration of study.
  Arms: Stage 1: PF-02417329 - Highest Dose
Drug: PF-04217329 - Vehicle — 1 drop of PF-04217329 vehicle, once a day, per dosed eye for duration of study.
  Arms: Stage 1: PF-04217329 - Vehicle
Drug: Latanoprost Vehicle — 1 drop of latanoprost vehicle, once a day, per dosed eye for duration of study.
  Arms: Stage 2: PF-04217329 - Low Dose + Latanoprost Vehicle
Drug: PF-04217329 - Low Dose — Five minutes after latanoprost vehicle, 1 drop of low dose PF-04217329, once a day, per dosed eye for duration of study.
  Arms: Stage 2: PF-04217329 - Low Dose + Latanoprost Vehicle
Drug: Latanoprost Vehicle — 1 drop of latanoprost vehicle, once a day, per dosed eye for duration of study.
  Arms: Stage 2: PF-04217329 - Middle Dose + Latanoprost Vehicle
Drug: PF-04217329 - Middle Dose — Five minutes after latanoprost vehicle, 1 drop of middle dose PF-04217329, once a day, per dosed eye for duration of study.
  Arms: Stage 2: PF-04217329 - Middle Dose + Latanoprost Vehicle
Drug: Latanoprost Vehicle — 1 drop of latanoprost vehicle, once a day, per dosed eye for duration of study.
  Arms: Stage 2: PF-04217329 - High Dose + Latanoprost Vehicle
Drug: PF-04217329 - High Dose — Five minutes after latanoprost vehicle, 1 drop of high dose PF-04217329, once a day, per dosed eye for duration of study.
  Arms: Stage 2: PF-04217329 - High Dose + Latanoprost Vehicle
Drug: Latanoprost 0.005% — 1 drop of latanoprost 0.005%, once a day, per dosed eye for duration of study.
  Arms: Stage 2: PF-04217329 - Low Dose + Latanoprost 0.005%
Drug: PF-04217329 - Low Dose — Five minutes after latanoprost 0.005%, 1 drop of low dose PF-04217329, once a day, per dosed eye for duration of study.
  Arms: Stage 2: PF-04217329 - Low Dose + Latanoprost 0.005%
Drug: Latanoprost 0.005% — 1 drop of latanoprost 0.005%, once a day, per dosed eye for duration of study.
  Arms: Stage 2: PF-04217329 - Middle Dose + Latanoprost 0.005%
Drug: PF-04217329 - Middle Dose — Five minutes after latanoprost 0.005%, 1 drop middle dose PF-04217329, once a day, per dosed eye for duration of study.
  Arms: Stage 2: PF-04217329 - Middle Dose + Latanoprost 0.005%
Drug: Latanoprost 0.005% — 1 drop of latanoprost 0.005%, once a day, per dosed eye for duration of study.
  Arms: Stage 2: PF-04217329 - High Dose + Latanoprost 0.005%
Drug: PF-04217329 - High Dose — Five minutes after latanoprost 0.005%, 1 drop high dose PF-04217329, once a day, per dosed eye for duration of study.
  Arms: Stage 2: PF-04217329 - High Dose + Latanoprost 0.005%
Drug: Latanoprost 0.005% — 1 drop of latanoprost 0.005%, once a day, per dosed eye for duration of study.
  Arms: Stage 2: PF-04217329 - Vehicle + Latanoprost 0.005%
Drug: PF-04217329 - Vehicle — Five minutes after latanoprost 0.005%, 1 drop of PF-04217329 vehicle, once a day, per dosed eye for duration of study.
  Arms: Stage 2: PF-04217329 - Vehicle + Latanoprost 0.005%

SUMMARY:
To evaluate the safety and efficacy of PF-04217329.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open-angle glaucoma (including pigmentary or pseudoexfoliative) or ocular hypertension in 1 or both eyes.
* Qualifying intraocular pressure (IOP) in the same eye at the Eligibility 1 and 2 measurements.

Exclusion Criteria:

* Closed/barely open anterior chamber angle or a history of acute angle closure in either eye.
* Anticipate the need to initiate or modify medication (systemic or topical) that is known to affect intraocular pressure (IOP) during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2007-12-11 (Actual); Primary Completion 2009-06-26 (Actual); Study Completion 2009-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- United States (23):
  - Sall Research Medical Center, Artesia, California
  - Eye Research Foundation, Newport Beach, California
  - North Bay Eye Associates, Inc., Petaluma, California
  - Centre For Health Care, Poway, California
  - Atlantic Institute of Clinical Research, Daytona Beach, Florida
  - Florida Health Care Plans, Daytona Beach, Florida
  - Eye Associates of Fort Myers, Fort Myers, Florida
  - International Eye Associates, PA, Ormond Beach, Florida
  - Coastal Research Associates,LLC, Atlanta, Georgia
  - Omni Eye Services of Atlanta, Atlanta, Georgia
  - Eye Care Centers Management, Inc., Morrow, Georgia
  - The Eye Group of Southern Indiana, Evansville, Indiana
  - Taustine Eye Center, Louisville, Kentucky
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - Charlotte Eye Ear Nose and Throat Associates, PA, Charlotte, North Carolina
  - Cornerstone Eye Care, High Point, North Carolina
  - Mark J. Weiss, MD. Inc., Tulsa, Oklahoma
  - Glaucoma Care Center at Century Eye Care, Bristol, Pennsylvania
  - Wills Eye Institute, Philadelphia, Pennsylvania
  - Bluestein Custom Vision, Charleston, South Carolina
  - Total Eye Care, PA, Memphis, Tennessee
  - Texan Eye Care, PA, Austin, Texas
  - Eye Physicians of Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Schachar RA, Raber S, Courtney R, Zhang M. A phase 2, randomized, dose-response trial of taprenepag isopropyl (PF-04217329) versus latanoprost 0.005% in open-angle glaucoma and ocular hypertension. Curr Eye Res. 2011 Sep;36(9):809-17. doi: 10.3109/02713683.2011.593725. PMID 21851167
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0191001&StudyName=Safety%20and%20efficacy%20of%20PF-04217329%20in%20patients%20with%20glaucoma%20or%20elevated%20eye%20pressure.

RESULTS

PARTICIPANT FLOW:
Groups:
- Taprenepag 0.0025% (Stage I): Participants self-administered 1 drop (27 microliter [mcL]) of taprenepag (taprenepag isopropyl, PF-04217329) 0.0025 percent (%) ophthalmic solution into each eye once daily for 14 days in Stage I.
- Taprenepag 0.005% (Stage I): Participants self-administered 1 drop (27 mcL) of taprenepag (taprenepag isopropyl, PF-04217329) 0.005% ophthalmic solution into each eye once daily for 14 days in Stage I.
- Taprenepag 0.01% (Stage I): Participants self-administered 1 drop (27 mcL) of taprenepag (taprenepag isopropyl, PF-04217329) 0.01% ophthalmic solution into each eye once daily for 14 days in Stage I.
- Taprenepag 0.015% (Stage I): Participants self-administered 1 drop (27 mcL) of taprenepag (taprenepag isopropyl, PF-04217329) 0.015% ophthalmic solution into each eye once daily for 14 days in Stage I.
- Taprenepag 0.02% (Stage I): Participants self-administered 1 drop (27 mcL) of taprenepag (taprenepag isopropyl, PF-04217329) 0.02% ophthalmic solution into each eye once daily for 14 days in Stage I.
- Taprenepag 0.03% (Stage I): Participants self-administered 1 drop (27 mcL) of taprenepag (taprenepag isopropyl, PF-04217329) 0.03% ophthalmic solution into each eye once daily for 14 days in Stage I.
- Taprenepag Vehicle (Stage I): Participants self-administered 1 drop (27 mcL) of vehicle matched to taprenepag (taprenepag isopropyl, PF-04217329) ophthalmic solution into each eye once daily for 14 days in Stage I.
- Latanoprost Vehicle and Taprenepag 0.005% (Stage II): Participants self-administered 1 drop (27 mcL) of vehicle matched to latanoprost ophthalmic solution followed by 1 drop (27 mcL) of taprenepag (taprenepag isopropyl, PF-04217329) 0.005% ophthalmic solution after 5 minutes, into each eye once daily for 28 days in Stage II.
- Latanoprost Vehicle and Taprenepag 0.01% (Stage II): Participants self-administered 1 drop (27 mcL) of vehicle matched to latanoprost ophthalmic solution followed by 1 drop (27 mcL) of taprenepag (taprenepag isopropyl, PF-04217329) 0.01% ophthalmic solution after 5 minutes, into each eye once daily for 28 days in Stage II.
- Latanoprost Vehicle and Taprenepag 0.015% (Stage II): Participants self-administered 1 drop (27 mcL) of vehicle matched to latanoprost ophthalmic solution followed by 1 drop (27 mcL) of taprenepag (taprenepag isopropyl, PF-04217329) 0.015% ophthalmic solution after 5 minutes, into each eye once daily for 28 days in Stage II.
- Latanoprost 0.005% and Taprenepag 0.005% (Stage II): Participants self-administered 1 drop (27 mcL) of latanoprost 0.005% ophthalmic solution followed by 1 drop (27 mcL) of taprenepag (taprenepag isopropyl, PF-04217329) 0.005% ophthalmic solution after 5 minutes, into each eye once daily for 28 days in Stage II.
- Latanoprost 0.005% and Taprenepag 0.01% (Stage II): Participants self-administered 1 drop (27 mcL) of latanoprost 0.005% ophthalmic solution followed by 1 drop (27 mcL) of taprenepag (taprenepag isopropyl, PF-04217329) 0.01% ophthalmic solution after 5 minutes, into each eye once daily for 28 days in Stage II.
- Latanoprost 0.005% and Taprenepag 0.015% (Stage II): Participants self-administered 1 drop (27 mcL) of latanoprost 0.005% ophthalmic solution followed by 1 drop (27 mcL) of taprenepag (taprenepag isopropyl, PF-04217329) 0.015% ophthalmic solution after 5 minutes, into each eye once daily for 28 days in Stage II.
- Latanoprost 0.005% and Taprenepag Vehicle (Stage II): Participants self-administered 1 drop (27 mcL) of latanoprost 0.005% ophthalmic solution followed by 1 drop (27 mcL) of vehicle matched to taprenepag (taprenepag isopropyl, PF-04217329) ophthalmic solution after 5 minutes, into each eye once daily for 28 days in Stage II.
Period: Stage I (14 Days)
Arm/Group | Taprenepag 0.0025% (Stage I) | Taprenepag 0.005% (Stage I) | Taprenepag 0.01% (Stage I) | Taprenepag 0.015% (Stage I) | Taprenepag 0.02% (Stage I) | Taprenepag 0.03% (Stage I) | Taprenepag Vehicle (Stage I) | Latanoprost Vehicle and Taprenepag 0.005% (Stage II) | Latanoprost Vehicle and Taprenepag 0.01% (Stage II) | Latanoprost Vehicle and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag 0.005% (Stage II) | Latanoprost 0.005% and Taprenepag 0.01% (Stage II) | Latanoprost 0.005% and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag Vehicle (Stage II)
Started | 9 | 9 | 9 | 10 | 9 | 9 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 9 | 9 | 9 | 10 | 8 | 6 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage II (28 Days)
Arm/Group | Taprenepag 0.0025% (Stage I) | Taprenepag 0.005% (Stage I) | Taprenepag 0.01% (Stage I) | Taprenepag 0.015% (Stage I) | Taprenepag 0.02% (Stage I) | Taprenepag 0.03% (Stage I) | Taprenepag Vehicle (Stage I) | Latanoprost Vehicle and Taprenepag 0.005% (Stage II) | Latanoprost Vehicle and Taprenepag 0.01% (Stage II) | Latanoprost Vehicle and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag 0.005% (Stage II) | Latanoprost 0.005% and Taprenepag 0.01% (Stage II) | Latanoprost 0.005% and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag Vehicle (Stage II)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 36 | 36 | 36 | 36 | 36 | 36
Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 36 | 36 | 36 | 36 | 36 | 35
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 33 | 33 | 31 | 32 | 31 | 34
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 5 | 4 | 5 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 4 | 5 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized, but not treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Taprenepag 0.0025% (Stage I) | Taprenepag 0.005% (Stage I) | Taprenepag 0.01% (Stage I) | Taprenepag 0.015% (Stage I) | Taprenepag 0.02% (Stage I) | Taprenepag 0.03% (Stage I) | Taprenepag Vehicle (Stage I) | Latanoprost Vehicle and Taprenepag 0.005% (Stage II) | Latanoprost Vehicle and Taprenepag 0.01% (Stage II) | Latanoprost Vehicle and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag 0.005% (Stage II) | Latanoprost 0.005% and Taprenepag 0.01% (Stage II) | Latanoprost 0.005% and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag Vehicle (Stage II) | Total
Number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 9 | 12 | 35 | 36 | 36 | 36 | 36 | 36 | 35 | 317
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (13.0) | 59.1 (8.1) | 64.1 (6.8) | 51.8 (10.4) | 64.6 (9.6) | 60.3 (8.5) | 62.1 (6.5) | 62.5 (10.7) | 63.8 (11.4) | 66.6 (10.1) | 66.7 (11.4) | 64.1 (9.1) | 63.7 (9.4) | 68.9 (10.2) | 64.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 6 | 10 | 3 | 6 | 8 | 25 | 22 | 21 | 24 | 25 | 21 | 22 | 204
  Male | 5 | 2 | 3 | 0 | 6 | 3 | 4 | 10 | 14 | 15 | 12 | 11 | 15 | 13 | 113

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Diurnal Intra Ocular Pressure (IOP) in Study Eye at Day 14: Stage I
Description: Diurnal IOP was defined as the mean IOP over 24 hours. IOP was measured using Goldmann applanation tonometer. IOP was measured in both the eyes, and the eye with higher IOP reading at the 2 eligibility visits was referred as 'study eye' for efficacy assessment. If both the measurements were equal, right eye was selected as the study eye. IOP was measured twice in the same eye, and if the difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), the mean of the 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline = diurnal IOP at baseline - diurnal IOP at Day 14.
Time Frame: Stage I: Baseline, Day 14
Population: ITT population included all randomized participants who received at least 1 dose of study medication. Last observation carried forward (LOCF) method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag 0.0025% (Stage I) | Taprenepag 0.005% (Stage I) | Taprenepag 0.01% (Stage I) | Taprenepag 0.015% (Stage I) | Taprenepag 0.02% (Stage I) | Taprenepag 0.03% (Stage I) | Taprenepag Vehicle (Stage I)
Number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 9 | 12
mmHg
  Baseline | 25.97 (2.420) | 26.25 (2.400) | 25.90 (2.094) | 26.44 (1.560) | 28.10 (3.102) | 26.26 (1.831) | 26.04 (2.182)
  Change at Day 14 | 3.65 (1.749) | 5.40 (2.508) | 7.18 (2.749) | 6.48 (4.278) | 6.00 (2.748) | 6.69 (4.563) | 0.64 (1.382)
Statistical Analysis 1: Comparison: Taprenepag 0.0025% (Stage I) vs Taprenepag Vehicle (Stage I); Analysis was based on analysis of covariance (ANCOVA) model for effect of taprenepag compared to its vehicle with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.028, ANCOVA; Least squares (LS) mean difference = 3.02, 90% CI 2-sided [0.78 to 5.25]
Statistical Analysis 2: Comparison: Taprenepag 0.005% (Stage I) vs Taprenepag Vehicle (Stage I); Analysis was based on ANCOVA model for effect of taprenepag compared to its vehicle with treatment and baseline IOP as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 4.73, 90% CI 2-sided [2.50 to 6.96]
Statistical Analysis 3: Comparison: Taprenepag 0.01% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.56, 90% CI 2-sided [4.33 to 8.79]
Statistical Analysis 4: Comparison: Taprenepag 0.015% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.78, 90% CI 2-sided [3.60 to 7.95]
Statistical Analysis 5: Comparison: Taprenepag 0.02% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.06, 90% CI 2-sided [2.74 to 7.37]
Statistical Analysis 6: Comparison: Taprenepag 0.03% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.02, 90% CI 2-sided [3.79 to 8.25]

2. Primary Outcome: Change From Baseline in Mean Diurnal Intra Ocular Pressure (IOP) in Study Eye at Day 28: Stage II
Description: Diurnal IOP was defined as the mean IOP over 24 hours. IOP was measured using Goldmann applanation tonometer. IOP was measured in both the eyes, and the eye with higher IOP reading at the 2 eligibility visits was referred as 'study eye' for efficacy assessment. If both the measurements were equal, right eye was selected as the study eye. IOP was measured twice in the same eye, and if the difference between 2 measurements was less than or equal to 2 mmHg, the mean of the 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline = diurnal IOP at baseline - diurnal IOP at Day 28.
Time Frame: Stage II: Baseline, Day 28
Population: ITT population included all randomized participants who received at least 1 dose of study medication. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Latanoprost Vehicle and Taprenepag 0.005% (Stage II) | Latanoprost Vehicle and Taprenepag 0.01% (Stage II) | Latanoprost Vehicle and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag 0.005% (Stage II) | Latanoprost 0.005% and Taprenepag 0.01% (Stage II) | Latanoprost 0.005% and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag Vehicle (Stage II)
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 36 | 36 | 35
mmHg
  Baseline | 25.75 (2.266) | 26.47 (2.563) | 26.69 (2.509) | 26.98 (2.813) | 26.36 (2.524) | 27.34 (2.876) | 26.81 (2.783)
  Change at Day 28 | 7.35 (3.559) | 7.05 (2.875) | 7.14 (3.462) | 8.29 (3.817) | 9.10 (3.292) | 8.78 (3.592) | 6.74 (2.927)
Statistical Analysis 1: Comparison: Latanoprost Vehicle and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.171, ANCOVA; LS mean difference = 1.06, 90% CI 2-sided [-0.21 to 2.32]
Statistical Analysis 2: Comparison: Latanoprost Vehicle and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.553, ANCOVA; LS mean difference = 0.45, 90% CI 2-sided [-0.80 to 1.70]
Statistical Analysis 3: Comparison: Latanoprost Vehicle and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.555, ANCOVA; LS mean difference = 0.45, 90% CI 2-sided [-0.80 to 1.70]
Statistical Analysis 4: Comparison: Latanoprost 0.005% and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Analysis was based on ANCOVA model for effect of taprenepag in combination with latanoprost compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.053, ANCOVA; LS mean difference = 1.48, 90% CI 2-sided [0.22 to 2.73]
Statistical Analysis 5: Comparison: Latanoprost 0.005% and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 2.54, 90% CI 2-sided [1.29 to 3.80]
Statistical Analysis 6: Comparison: Latanoprost 0.005% and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.018, ANCOVA; LS mean difference = 1.81, 90% CI 2-sided [0.56 to 3.07]

3. Primary Outcome: Number of Participants With Treatment Emergent Ocular Adverse Events (AEs): Stage I
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study medication and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Ocular AEs were the events which were localized in the ocular region.
Time Frame: Stage I: Day 1 up to 28 days after last dose of study medication (up to 44 days)
Population: ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Taprenepag 0.0025% (Stage I) | Taprenepag 0.005% (Stage I) | Taprenepag 0.01% (Stage I) | Taprenepag 0.015% (Stage I) | Taprenepag 0.02% (Stage I) | Taprenepag 0.03% (Stage I) | Taprenepag Vehicle (Stage I)
Number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 9 | 12
Participants | 1 | 2 | 0 | 5 | 4 | 9 | 3

4. Primary Outcome: Number of Participants With Treatment Emergent Ocular Adverse Events (AEs): Stage II
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study medication and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Ocular AEs were the events which were localized in the ocular region.
Time Frame: Stage II: Day 1 up to 28 days after last dose of study medication (up to 59 days)
Population: ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Latanoprost Vehicle and Taprenepag 0.005% (Stage II) | Latanoprost Vehicle and Taprenepag 0.01% (Stage II) | Latanoprost Vehicle and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag 0.005% (Stage II) | Latanoprost 0.005% and Taprenepag 0.01% (Stage II) | Latanoprost 0.005% and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag Vehicle (Stage II)
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 36 | 36 | 35
Participants | 17 | 20 | 27 | 24 | 26 | 26 | 14

5. Secondary Outcome: Mean Intra Ocular Pressure (IOP) in Study Eye: Stage I
Description: IOP was measured using Goldmann applanation tonometer. IOP was measured in both the eyes, and the eye with higher IOP reading at the 2 eligibility visits was referred as 'study eye' for efficacy assessment. If both the measurements were equal, right eye was selected as the study eye. IOP was measured twice in the same eye, and if the difference between 2 measurements was less than or equal to 2 mmHg, the mean of the 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values.
Time Frame: Stage I: 8 ante meridiem (AM) on Day 1, 8 AM, 10 AM, 1 post meridiem (PM), 4 PM on Day 7, and 14
Population: ITT population included all randomized participants who received at least 1 dose of study medication. LOCF method was used to impute missing values. Here 'number analyzed' signifies participants evaluable each specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag 0.0025% (Stage I) | Taprenepag 0.005% (Stage I) | Taprenepag 0.01% (Stage I) | Taprenepag 0.015% (Stage I) | Taprenepag 0.02% (Stage I) | Taprenepag 0.03% (Stage I) | Taprenepag Vehicle (Stage I)
Number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 9 | 12
mmHg
  Day 1: 8 AM | 22.89 (3.140) | 22.28 (3.709) | 20.00 (1.677) | 21.70 (3.425) | 22.06 (2.732) | 21.22 (4.214) | 26.79 (4.335)
  Day 7: 8 AM | 23.22 (3.563) | 21.06 (2.888) | 19.44 (4.081) | 20.25 (4.584) | 20.22 (3.866) | 20.78 (3.420) | 26.00 (4.843)
  Day 7: 10 AM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 8 | 8 | 12
  Day 7: 10 AM | 21.17 (2.165) | 19.11 (3.943) | 18.39 (3.110) | 19.15 (4.429) | 20.38 (2.888) | 17.44 (3.803) | 25.46 (4.293)
  Day 7: 1 PM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 8 | 8 | 12
  Day 7: 1 PM | 21.17 (2.525) | 19.83 (3.269) | 17.22 (4.063) | 17.55 (3.905) | 20.63 (4.224) | 18.25 (4.359) | 23.63 (2.909)
  Day 7: 4 PM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 8 | 8 | 12
  Day 7: 4 PM | 21.17 (3.491) | 20.06 (5.282) | 17.61 (3.935) | 16.95 (3.954) | 20.88 (4.604) | 18.63 (3.926) | 25.58 (5.044)
  Day 14: 8 AM | 24.33 (4.737) | 21.61 (3.927) | 19.28 (2.438) | 20.75 (4.906) | 22.94 (3.787) | 20.17 (5.750) | 26.58 (4.592)
  Day 14: 10 AM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 8 | 12
  Day 14: 10 AM | 20.89 (1.635) | 19.78 (2.740) | 18.28 (3.501) | 19.90 (4.858) | 21.89 (3.798) | 18.06 (4.724) | 24.46 (2.463)
  Day 14: 1 PM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 8 | 12
  Day 14: 1 PM | 21.28 (2.078) | 20.83 (2.839) | 18.56 (3.754) | 19.60 (5.254) | 22.89 (4.029) | 18.50 (3.703) | 25.46 (3.665)
  Day 14: 4 PM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 8 | 12
  Day 14: 4 PM | 22.78 (3.914) | 21.17 (3.841) | 18.78 (3.970) | 19.60 (5.004) | 20.67 (2.704) | 19.06 (3.886) | 25.08 (3.154)

6. Secondary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 1 (8 AM), 7 and 14 (8 AM, 10 AM, 1 PM, 4 PM): Stage I
Description: IOP was measured using Goldmann applanation tonometer. IOP was measured in both eyes, and the eye with higher IOP reading at 2 eligibility visits was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as the study eye. IOP was measured twice in the same eye, and if the difference between 2 measurements was less than or equal to 2 mmHg, the mean of the 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline = baseline IOP - post-baseline IOP. Change at various post-dose time points was calculated from the baseline values at same time points on Day 0 (for example, value at 8 AM on Day 0 was used as baseline value for 8 AM value on Day 1, 7 and 14).
Time Frame: Stage I: 8 AM, 10 AM, 1 PM, 4 PM on Day 0 (Baseline), 8 AM on Day 1, 8 AM, 10 AM, 1 PM, 4 PM on Day 7, and 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag 0.0025% (Stage I) | Taprenepag 0.005% (Stage I) | Taprenepag 0.01% (Stage I) | Taprenepag 0.015% (Stage I) | Taprenepag 0.02% (Stage I) | Taprenepag 0.03% (Stage I) | Taprenepag Vehicle (Stage I)
Number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 9 | 12
mmHg
  Day0: Baseline for Day 1, 7, 14 8 AM | 27.78 (1.847) | 27.72 (1.693) | 27.72 (2.403) | 28.45 (1.471) | 29.81 (2.769) | 28.44 (1.887) | 28.15 (2.625)
  Day 0: Baseline for Day 7 10 AM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 8 | 8 | 12
  Day 0: Baseline for Day 7 10 AM | 24.75 (1.916) | 26.11 (2.494) | 25.94 (2.872) | 26.30 (1.285) | 26.53 (1.906) | 26.16 (2.507) | 25.13 (2.519)
  Day 0: Baseline for Day 7 1 PM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 8 | 8 | 12
  Day 0: Baseline for Day 7 1 PM | 25.83 (3.279) | 26.06 (2.965) | 25.08 (2.208) | 25.10 (2.289) | 27.13 (3.009) | 25.69 (2.191) | 25.52 (2.742)
  Day 0: Baseline for Day 7 4 PM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 8 | 8 | 12
  Day 0: Baseline for Day 7 4 PM | 25.50 (3.403) | 25.11 (3.113) | 24.86 (2.405) | 25.90 (2.237) | 26.41 (3.068) | 25.28 (1.925) | 25.35 (2.907)
  Day 0:Baseline for Day 14 10 AM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 8 | 12
  Day 0:Baseline for Day 14 10 AM | 24.75 (1.916) | 26.11 (2.494) | 25.94 (2.872) | 26.30 (1.285) | 27.44 (3.269) | 26.16 (2.507) | 25.13 (2.519)
  Day 0:Baseline for Day 14 1 PM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 8 | 12
  Day 0:Baseline for Day 14 1 PM | 25.83 (3.279) | 26.06 (2.965) | 25.08 (2.208) | 25.10 (2.289) | 28.03 (3.906) | 25.69 (2.191) | 25.52 (2.742)
  Day 0:Baseline for Day 14 4 PM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 8 | 12
  Day 0:Baseline for Day 14 4 PM | 25.50 (3.403) | 25.11 (3.113) | 24.86 (2.405) | 25.90 (2.237) | 27.11 (3.564) | 25.28 (1.925) | 25.35 (2.907)
  Change at Day 1 8 AM | 4.89 (2.302) | 5.44 (3.154) | 7.72 (2.697) | 6.75 (2.875) | 7.75 (3.276) | 7.22 (4.459) | 1.35 (2.702)
  Change at Day 7 8 AM | 4.56 (2.957) | 6.67 (1.644) | 8.28 (4.186) | 8.20 (3.885) | 9.58 (3.356) | 7.67 (4.373) | 2.15 (3.224)
  Change at Day 7 10 AM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 8 | 8 | 12
  Change at Day 7 10 AM | 3.58 (3.064) | 7.00 (3.219) | 7.56 (3.041) | 7.15 (4.301) | 6.16 (2.891) | 8.72 (4.137) | -0.33 (3.099)
  Change at Day 7 1 PM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 8 | 8 | 12
  Change at Day 7 1 PM | 4.67 (3.255) | 6.22 (2.498) | 7.86 (2.908) | 7.55 (3.947) | 6.50 (4.652) | 7.44 (3.351) | 1.90 (2.546)
  Change at Day 7 4 PM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 8 | 8 | 12
  Change at Day 7 4 PM | 4.33 (2.880) | 5.06 (4.083) | 7.25 (2.929) | 8.95 (3.787) | 5.53 (4.519) | 6.66 (3.744) | -0.23 (2.940)
  Change at Day 14 8 AM | 3.44 (3.964) | 6.11 (3.518) | 8.44 (2.267) | 7.70 (3.994) | 6.86 (2.622) | 8.28 (5.701) | 1.56 (2.962)
  Change at Day 14 10 AM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 8 | 12
  Change at Day 14 10 AM | 3.86 (1.768) | 6.33 (2.559) | 7.67 (3.245) | 6.40 (4.754) | 5.56 (3.273) | 8.09 (4.274) | 0.67 (3.085)
  Change at Day 14 1 PM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 8 | 12
  Change at Day 14 1 PM | 4.56 (2.524) | 5.22 (2.673) | 6.53 (2.746) | 5.50 (4.419) | 5.14 (3.664) | 7.19 (2.930) | 0.06 (2.794)
  Change at Day 14 4 PM: number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 8 | 12
  Change at Day 14 4 PM | 2.72 (1.950) | 3.94 (2.880) | 6.08 (3.573) | 6.30 (5.296) | 6.44 (3.015) | 6.22 (4.021) | 0.27 (1.804)
Statistical Analysis 1: Comparison: Taprenepag 0.0025% (Stage I) vs Taprenepag Vehicle (Stage I); Change at Day 1 8 AM: Analysis was based on ANCOVA model for effect of taprenepag compared to its vehicle with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.011, ANCOVA; LS mean difference = 3.62, 90% CI 2-sided [1.34 to 5.90]
Statistical Analysis 2: Comparison: Taprenepag 0.005% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.004, ANCOVA; LS mean difference = 4.19, 90% CI 2-sided [1.91 to 6.47]
Statistical Analysis 3: Comparison: Taprenepag 0.01% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.47, 90% CI 2-sided [4.19 to 8.75]
Statistical Analysis 4: Comparison: Taprenepag 0.015% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.32, 90% CI 2-sided [3.11 to 7.54]
Statistical Analysis 5: Comparison: Taprenepag 0.02% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.00, 90% CI 2-sided [3.66 to 8.33]
Statistical Analysis 6: Comparison: Taprenepag 0.03% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.80, 90% CI 2-sided [3.52 to 8.08]
Statistical Analysis 7: Comparison: Taprenepag 0.0025% (Stage I) vs Taprenepag Vehicle (Stage I); Change at Day 7 8 AM: Analysis was based on ANCOVA model for effect of taprenepag compared to its vehicle with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.120, ANCOVA; LS mean difference = 2.44, 90% CI 2-sided [-0.14 to 5.02]
Statistical Analysis 8: Comparison: Taprenepag 0.005% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.005, ANCOVA; LS mean difference = 4.55, 90% CI 2-sided [1.97 to 7.14]
Statistical Analysis 9: Comparison: Taprenepag 0.01% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.17, 90% CI 2-sided [3.58 to 8.75]
Statistical Analysis 10: Comparison: Taprenepag 0.015% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.03, 90% CI 2-sided [3.52 to 8.54]
Statistical Analysis 11: Comparison: Taprenepag 0.02% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 7.31, 90% CI 2-sided [4.66 to 9.95]
Statistical Analysis 12: Comparison: Taprenepag 0.03% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.50, 90% CI 2-sided [2.91 to 8.08]
Statistical Analysis 13: Comparison: Taprenepag 0.0025% (Stage I) vs Taprenepag Vehicle (Stage I); Change at Day 7 10 AM: Analysis was based on ANCOVA model for effect of taprenepag compared to its vehicle with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.009, ANCOVA; LS mean difference = 4.04, 90% CI 2-sided [1.56 to 6.53]
Statistical Analysis 14: Comparison: Taprenepag 0.005% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 7.00, 90% CI 2-sided [4.49 to 9.50]
Statistical Analysis 15: Comparison: Taprenepag 0.01% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 7.61, 90% CI 2-sided [5.11 to 10.11]
Statistical Analysis 16: Comparison: Taprenepag 0.015% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 7.08, 90% CI 2-sided [4.64 to 9.53]
Statistical Analysis 17: Comparison: Taprenepag 0.02% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.01, 90% CI 2-sided [3.40 to 8.62]
Statistical Analysis 18: Comparison: Taprenepag 0.03% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 8.70, 90% CI 2-sided [6.11 to 11.30]
Statistical Analysis 19: Comparison: Taprenepag 0.0025% (Stage I) vs Taprenepag Vehicle (Stage I); Change at Day 7 1 PM: Analysis was based on ANCOVA model for effect of taprenepag compared to its vehicle with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.066, ANCOVA; LS mean difference = 2.66, 90% CI 2-sided [0.29 to 5.02]
Statistical Analysis 20: Comparison: Taprenepag 0.005% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; p = 0.006, ANCOVA; LS mean difference = 4.13, 90% CI 2-sided [1.76 to 6.50]
Statistical Analysis 21: Comparison: Taprenepag 0.01% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.13, 90% CI 2-sided [3.76 to 8.49]
Statistical Analysis 22: Comparison: Taprenepag 0.015% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.81, 90% CI 2-sided [3.51 to 8.11]
Statistical Analysis 23: Comparison: Taprenepag 0.02% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; p = 0.010, ANCOVA; LS mean difference = 4.02, 90% CI 2-sided [1.53 to 6.50]
Statistical Analysis 24: Comparison: Taprenepag 0.03% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.48, 90% CI 2-sided [3.03 to 7.93]
Statistical Analysis 25: Comparison: Taprenepag 0.0025% (Stage I) vs Taprenepag Vehicle (Stage I); Change at Day 7 4 PM: Analysis was based on ANCOVA model for effect of taprenepag compared to its vehicle with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.006, ANCOVA; LS mean difference = 4.55, 90% CI 2-sided [1.91 to 7.19]
Statistical Analysis 26: Comparison: Taprenepag 0.005% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS mean difference = 5.30, 90% CI 2-sided [2.66 to 7.94]
Statistical Analysis 27: Comparison: Taprenepag 0.01% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 7.51, 90% CI 2-sided [4.87 to 10.16]
Statistical Analysis 28: Comparison: Taprenepag 0.015% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 9.14, 90% CI 2-sided [6.57 to 11.71]
Statistical Analysis 29: Comparison: Taprenepag 0.02% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS mean difference = 5.69, 90% CI 2-sided [2.94 to 8.44]
Statistical Analysis 30: Comparison: Taprenepag 0.03% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.89, 90% CI 2-sided [4.16 to 9.62]
Statistical Analysis 31: Comparison: Taprenepag 0.0025% (Stage I) vs Taprenepag Vehicle (Stage I); Change at Day 14 8 AM: Analysis was based on ANCOVA model for effect of taprenepag compared to its vehicle with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.269, ANCOVA; LS mean difference = 1.83, 90% CI 2-sided [-0.91 to 4.58]
Statistical Analysis 32: Comparison: Taprenepag 0.005% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 31]; Test type: Superiority or Other; p = 0.009, ANCOVA; LS mean difference = 4.49, 90% CI 2-sided [1.75 to 7.24]
Statistical Analysis 33: Comparison: Taprenepag 0.01% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 31]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.83, 90% CI 2-sided [4.08 to 9.57]
Statistical Analysis 34: Comparison: Taprenepag 0.015% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 31]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.18, 90% CI 2-sided [3.52 to 8.84]
Statistical Analysis 35: Comparison: Taprenepag 0.02% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 31]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS mean difference = 5.52, 90% CI 2-sided [2.71 to 8.33]
Statistical Analysis 36: Comparison: Taprenepag 0.03% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 31]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.76, 90% CI 2-sided [4.01 to 9.50]
Statistical Analysis 37: Comparison: Taprenepag 0.0025% (Stage I) vs Taprenepag Vehicle (Stage I); Change at Day 14 10 AM: Analysis was based on ANCOVA model for effect of taprenepag compared to its vehicle with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.024, ANCOVA; LS mean difference = 3.36, 90% CI 2-sided [0.95 to 5.76]
Statistical Analysis 38: Comparison: Taprenepag 0.005% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 37]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.24, 90% CI 2-sided [2.82 to 7.66]
Statistical Analysis 39: Comparison: Taprenepag 0.01% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 37]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.64, 90% CI 2-sided [4.23 to 9.06]
Statistical Analysis 40: Comparison: Taprenepag 0.015% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 37]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.22, 90% CI 2-sided [2.87 to 7.58]
Statistical Analysis 41: Comparison: Taprenepag 0.02% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 37]; Test type: Superiority or Other; p = 0.012, ANCOVA; LS mean difference = 3.88, 90% CI 2-sided [1.39 to 6.37]
Statistical Analysis 42: Comparison: Taprenepag 0.03% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 37]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.98, 90% CI 2-sided [4.48 to 9.48]
Statistical Analysis 43: Comparison: Taprenepag 0.0025% (Stage I) vs Taprenepag 0.005% (Stage I); Change at Day 14 1 PM: Analysis was based on ANCOVA model for effect of taprenepag compared to its vehicle with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.003, ANCOVA; LS mean difference = 4.41, 90% CI 2-sided [2.11 to 6.72]
Statistical Analysis 44: Comparison: Taprenepag 0.005% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 43]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.02, 90% CI 2-sided [2.72 to 7.33]
Statistical Analysis 45: Comparison: Taprenepag 0.01% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 43]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 6.58, 90% CI 2-sided [4.27 to 8.88]
Statistical Analysis 46: Comparison: Taprenepag 0.015% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 43]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.54, 90% CI 2-sided [3.31 to 7.78]
Statistical Analysis 47: Comparison: Taprenepag 0.02% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 43]; Test type: Superiority or Other; p = 0.003, ANCOVA; LS mean difference = 4.44, 90% CI 2-sided [2.06 to 6.82]
Statistical Analysis 48: Comparison: Taprenepag 0.03% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 43]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 7.08, 90% CI 2-sided [4.70 to 9.47]
Statistical Analysis 49: Comparison: Taprenepag 0.0025% (Stage I) vs Taprenepag Vehicle (Stage I); Change at Day 14 4 PM: Analysis was based on ANCOVA model for effect of taprenepag compared to its vehicle with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.103, ANCOVA; LS mean difference = 2.41, 90% CI 2-sided [-0.02 to 4.84]
Statistical Analysis 50: Comparison: Taprenepag 0.005% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 49]; Test type: Superiority or Other; p = 0.013, ANCOVA; LS mean difference = 3.75, 90% CI 2-sided [1.32 to 6.18]
Statistical Analysis 51: Comparison: Taprenepag 0.01% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.96, 90% CI 2-sided [3.53 to 8.39]
Statistical Analysis 52: Comparison: Taprenepag 0.015% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.87, 90% CI 2-sided [3.50 to 8.23]
Statistical Analysis 53: Comparison: Taprenepag 0.02% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.65, 90% CI 2-sided [3.18 to 8.11]
Statistical Analysis 54: Comparison: Taprenepag 0.03% (Stage I) vs Taprenepag Vehicle (Stage I); [analysis description as in outcome 6, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 5.97, 90% CI 2-sided [3.46 to 8.48]

7. Secondary Outcome: Mean Intra Ocular Pressure (IOP) in Study Eye: Stage II
Description: as for outcome 5
Time Frame: Stage II: 8 AM on Day 1; 8 AM, 10 AM, 1 PM, 4 PM on Days 7, 14, and 28
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Latanoprost Vehicle and Taprenepag 0.005% (Stage II) | Latanoprost Vehicle and Taprenepag 0.01% (Stage II) | Latanoprost Vehicle and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag 0.005% (Stage II) | Latanoprost 0.005% and Taprenepag 0.01% (Stage II) | Latanoprost 0.005% and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag Vehicle (Stage II)
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 36 | 36 | 35
mmHg
  Day 1: 8 AM: number analyzed (Participants) | 34 | 35 | 36 | 35 | 36 | 36 | 33
  Day 1: 8 AM | 19.12 (3.514) | 21.91 (3.177) | 20.61 (2.859) | 19.39 (3.229) | 18.76 (4.058) | 19.69 (3.945) | 20.39 (3.548)
  Day 7: 8 AM | 18.34 (3.115) | 19.40 (3.308) | 19.68 (3.140) | 18.83 (2.908) | 17.41 (4.035) | 18.28 (3.718) | 20.10 (3.698)
  Day 7: 10 AM: number analyzed (Participants) | 34 | 36 | 33 | 30 | 33 | 32 | 35
  Day 7: 10 AM | 17.26 (2.456) | 18.96 (3.938) | 18.61 (2.814) | 17.94 (2.551) | 16.80 (4.670) | 17.34 (3.028) | 19.10 (3.727)
  Day 7: 1 PM: number analyzed (Participants) | 34 | 36 | 33 | 30 | 33 | 32 | 35
  Day 7: 1 PM | 17.25 (3.184) | 18.68 (3.122) | 18.73 (3.518) | 18.02 (2.872) | 16.80 (4.219) | 17.09 (3.057) | 19.30 (3.032)
  Day 7: 4 PM: number analyzed (Participants) | 34 | 36 | 33 | 30 | 33 | 32 | 35
  Day 7: 4 PM | 17.26 (2.962) | 18.67 (3.690) | 18.27 (3.047) | 17.65 (2.998) | 16.91 (4.320) | 17.56 (2.989) | 19.70 (3.642)
  Day 14: 8 AM | 18.85 (3.439) | 19.56 (3.288) | 19.72 (3.644) | 19.53 (3.572) | 17.69 (4.580) | 18.67 (4.127) | 19.66 (3.908)
  Day 14: 10 AM: number analyzed (Participants) | 35 | 36 | 35 | 33 | 33 | 33 | 35
  Day 14: 10 AM | 17.81 (3.848) | 19.61 (4.209) | 19.44 (3.318) | 18.98 (3.318) | 16.66 (4.743) | 17.85 (3.282) | 19.40 (3.485)
  Day 14: 1 PM: number analyzed (Participants) | 35 | 36 | 35 | 33 | 33 | 33 | 35
  Day 14: 1 PM | 17.94 (3.912) | 19.33 (3.619) | 18.96 (3.776) | 18.89 (3.219) | 16.52 (4.622) | 17.35 (2.612) | 18.83 (3.231)
  Day 14: 4 PM: number analyzed (Participants) | 35 | 36 | 35 | 32 | 33 | 33 | 35
  Day 14: 4 PM | 17.41 (3.452) | 19.35 (4.035) | 18.31 (3.370) | 18.66 (3.117) | 16.98 (5.077) | 18.26 (2.736) | 19.54 (3.361)
  Day 28: 8 AM | 19.60 (3.794) | 19.76 (3.188) | 20.28 (4.294) | 19.11 (3.280) | 17.97 (4.876) | 18.99 (3.644) | 20.69 (3.577)
  Day 28: 10 AM: number analyzed (Participants) | 35 | 36 | 35 | 34 | 33 | 33 | 35
  Day 28: 10 AM | 17.93 (3.341) | 19.44 (3.335) | 19.74 (3.764) | 18.38 (3.038) | 16.86 (4.827) | 17.67 (3.196) | 19.64 (3.966)
  Day 28: 1 PM: number analyzed (Participants) | 35 | 36 | 35 | 34 | 33 | 33 | 35
  Day 28: 1 PM | 18.30 (3.787) | 19.19 (3.092) | 19.06 (3.399) | 18.47 (2.396) | 16.68 (5.331) | 17.39 (2.680) | 19.33 (3.204)
  Day 28: 4 PM: number analyzed (Participants) | 35 | 36 | 35 | 33 | 33 | 33 | 35
  Day 28: 4 PM | 17.79 (3.673) | 19.08 (3.394) | 19.13 (4.396) | 19.06 (2.772) | 17.12 (4.823) | 18.56 (3.323) | 20.06 (3.668)

8. Secondary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 1 (8 AM), 7 (8 AM, 10 AM, 1 PM, 4 PM), 14 (8 AM, 10 AM, 1 PM, 4 PM) and Day 28 (8 AM, 10 AM, 1 PM, 4 PM): Stage II
Description: IOP was measured using Goldmann applanation tonometer. IOP was measured in both eyes, and the eye with higher IOP reading at 2 eligibility visits was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as the study eye. IOP was measured twice in the same eye, and if the difference between 2 measurements was less than or equal to 2 mmHg, the mean of the 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline = baseline IOP - post-baseline IOP. Change at various post-dose time points was calculated from the baseline values at same time points on Day 0 (for example, value at 8 AM on Day 0 was used as baseline value for 8 AM value on Day 1, 7, 14 and 28).
Time Frame: Stage II: 8 AM, 10 AM, 1 PM, and 4 PM on Day 0 (Baseline), 8 AM on Day 1; 8 AM, 10 AM, 1 PM, 4 PM on Days 7, 14, and 28
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Latanoprost Vehicle and Taprenepag 0.005% (Stage II) | Latanoprost Vehicle and Taprenepag 0.01% (Stage II) | Latanoprost Vehicle and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag 0.005% (Stage II) | Latanoprost 0.005% and Taprenepag 0.01% (Stage II) | Latanoprost 0.005% and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag Vehicle (Stage II)
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 36 | 36 | 35
mmHg
  Day 0: Baseline for Day 1: 8AM: number analyzed (Participants) | 34 | 35 | 36 | 35 | 36 | 36 | 33
  Day 0: Baseline for Day 1: 8AM | 27.34 (1.525) | 28.21 (2.349) | 28.27 (2.155) | 29.10 (2.714) | 28.63 (2.648) | 29.19 (2.962) | 28.55 (2.728)
  Day 0: Baseline for Day 7,14,28: 8AM | 27.59 (2.098) | 28.16 (2.333) | 28.27 (2.155) | 29.03 (2.710) | 28.63 (2.648) | 29.19 (2.962) | 28.60 (2.656)
  Day 0: Baseline for Day 7: 10AM: number analyzed (Participants) | 34 | 36 | 33 | 30 | 33 | 32 | 35
  Day 0: Baseline for Day 7: 10AM | 25.74 (3.129) | 26.44 (3.005) | 26.70 (2.937) | 27.13 (3.453) | 26.42 (2.779) | 27.48 (3.450) | 26.70 (3.250)
  Day 0: Baseline for Day 7: 1PM: number analyzed (Participants) | 34 | 36 | 33 | 30 | 33 | 32 | 35
  Day 0: Baseline for Day 7: 1PM | 24.85 (2.501) | 25.67 (2.754) | 26.19 (2.992) | 26.04 (3.179) | 25.34 (2.707) | 26.27 (3.335) | 25.99 (2.863)
  Day 0: Baseline for Day 7: 4PM: number analyzed (Participants) | 34 | 36 | 33 | 30 | 33 | 32 | 35
  Day 0: Baseline for Day 7: 4PM | 24.83 (2.901) | 25.59 (3.040) | 25.87 (3.054) | 25.92 (3.293) | 25.35 (3.117) | 26.12 (3.154) | 25.84 (3.243)
  Day 0: Baseline for Day 14: 10AM: number analyzed (Participants) | 35 | 36 | 35 | 33 | 33 | 33 | 35
  Day 0: Baseline for Day 14: 10AM | 25.70 (3.089) | 26.44 (3.005) | 26.66 (2.854) | 26.94 (3.449) | 26.42 (2.779) | 27.41 (3.423) | 26.70 (3.250)
  Day 0: Baseline for Day 14: 1PM: number analyzed (Participants) | 35 | 36 | 35 | 33 | 33 | 33 | 35
  Day 0: Baseline for Day 14: 1PM | 24.84 (2.466) | 25.67 (2.754) | 26.13 (2.949) | 25.92 (3.068) | 25.34 (2.707) | 26.21 (3.297) | 25.99 (2.863)
  Day 0: Baseline for Day 14: 4PM: number analyzed (Participants) | 35 | 36 | 35 | 32 | 33 | 33 | 35
  Day 0: Baseline for Day 14: 4PM | 24.87 (2.868) | 25.59 (3.040) | 25.86 (3.013) | 25.99 (3.206) | 25.35 (3.117) | 26.20 (3.145) | 25.84 (3.243)
  Day 0: Baseline for Day 28: 10AM: number analyzed (Participants) | 35 | 36 | 35 | 34 | 33 | 33 | 35
  Day 0: Baseline for Day 28: 10AM | 25.70 (3.089) | 26.44 (3.005) | 26.66 (2.854) | 27.06 (3.467) | 26.42 (2.779) | 27.41 (3.423) | 26.70 (3.250)
  Day 0: Baseline for Day 28: 1PM: number analyzed (Participants) | 35 | 36 | 35 | 34 | 33 | 33 | 35
  Day 0: Baseline for Day 28: 1PM | 24.84 (2.466) | 25.67 (2.754) | 26.13 (2.949) | 25.98 (3.042) | 25.34 (2.707) | 26.21 (3.297) | 25.99 (2.863)
  Day 0: Baseline for Day 28: 4PM: number analyzed (Participants) | 35 | 36 | 35 | 33 | 33 | 33 | 35
  Day 0: Baseline for Day 28: 4PM | 24.87 (2.868) | 25.59 (3.040) | 25.86 (3.013) | 26.00 (3.156) | 25.35 (3.117) | 26.20 (3.145) | 25.84 (3.243)
  Change at Day 1: 8AM: number analyzed (Participants) | 34 | 35 | 36 | 35 | 36 | 36 | 33
  Change at Day 1: 8AM | 8.22 (4.071) | 6.29 (3.117) | 7.66 (3.110) | 9.72 (3.484) | 9.87 (2.786) | 9.49 (4.242) | 8.16 (4.031)
  Change at Day 7: 8AM | 9.24 (3.987) | 8.76 (3.459) | 8.59 (3.317) | 10.20 (3.497) | 11.22 (3.393) | 10.91 (3.623) | 8.50 (3.343)
  Change at Day 7: 10AM: number analyzed (Participants) | 34 | 36 | 33 | 30 | 33 | 32 | 35
  Change at Day 7: 10AM | 8.47 (3.754) | 7.49 (3.057) | 8.10 (3.328) | 9.19 (3.646) | 9.61 (3.448) | 10.14 (2.935) | 7.60 (3.031)
  Change at Day 7: 1PM: number analyzed (Participants) | 34 | 36 | 33 | 30 | 33 | 32 | 35
  Change at Day 7: 1PM | 7.60 (3.499) | 6.99 (2.943) | 7.46 (3.576) | 8.02 (4.046) | 8.54 (3.043) | 9.17 (4.022) | 6.69 (2.996)
  Change at Day 7: 4PM: number analyzed (Participants) | 34 | 36 | 33 | 30 | 33 | 32 | 35
  Change at Day 7: 4PM | 7.57 (3.525) | 6.92 (3.552) | 7.60 (3.388) | 8.27 (3.161) | 8.44 (2.888) | 8.55 (3.081) | 6.14 (3.011)
  Change at Day 14: 8AM | 8.74 (3.829) | 8.60 (3.254) | 8.55 (3.473) | 9.50 (3.915) | 10.94 (3.793) | 10.52 (4.446) | 8.94 (3.462)
  Change at Day 14: 10AM: number analyzed (Participants) | 35 | 36 | 35 | 33 | 33 | 33 | 35
  Change at Day 14: 10AM | 7.89 (4.568) | 6.83 (3.151) | 7.22 (3.292) | 7.95 (3.900) | 9.76 (3.467) | 9.56 (3.121) | 7.30 (2.397)
  Change at Day 14: 1PM: number analyzed (Participants) | 35 | 36 | 35 | 33 | 33 | 33 | 35
  Change at Day 14: 1PM | 6.89 (4.225) | 6.33 (2.837) | 7.17 (3.502) | 7.03 (3.710) | 8.83 (3.364) | 8.86 (3.710) | 7.16 (3.229)
  Change at Day 14: 4PM: number analyzed (Participants) | 35 | 36 | 35 | 32 | 33 | 33 | 35
  Change at Day 14: 4PM | 7.46 (3.725) | 6.24 (3.510) | 7.55 (3.392) | 7.33 (3.649) | 8.36 (3.721) | 7.95 (3.045) | 6.30 (3.746)
  Change at Day 28: 8AM | 7.99 (4.108) | 8.40 (3.501) | 8.00 (3.851) | 9.92 (3.845) | 10.66 (3.741) | 10.20 (3.958) | 7.91 (2.802)
  Change at Day 28: 10AM: number analyzed (Participants) | 35 | 36 | 35 | 34 | 33 | 33 | 35
  Change at Day 28: 10AM | 7.78 (3.987) | 7.00 (3.383) | 6.92 (3.706) | 8.68 (4.674) | 9.55 (3.561) | 9.74 (3.743) | 7.06 (3.311)
  Change at Day 28: 1PM: number analyzed (Participants) | 35 | 36 | 35 | 34 | 33 | 33 | 35
  Change at Day 28: 1PM | 6.54 (3.965) | 6.47 (2.645) | 7.07 (3.472) | 7.51 (3.915) | 8.66 (4.073) | 8.82 (4.037) | 6.66 (2.804)
  Change at Day 28: 4PM: number analyzed (Participants) | 35 | 36 | 35 | 33 | 33 | 33 | 35
  Change at Day 28: 4PM | 7.09 (3.938) | 6.51 (3.302) | 6.74 (4.480) | 6.94 (3.962) | 8.23 (3.420) | 7.64 (3.762) | 5.79 (3.219)
Statistical Analysis 1: Comparison: Latanoprost Vehicle and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 1 8 AM: Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.377, ANCOVA; LS mean difference = 0.72, 90% CI 2-sided [-0.63 to 2.08]
Statistical Analysis 2: Comparison: Latanoprost Vehicle and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.039, ANCOVA; LS mean difference = -1.68, 90% CI 2-sided [-3.01 to -0.35]
Statistical Analysis 3: Comparison: Latanoprost Vehicle and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.668, ANCOVA; LS mean difference = -0.34, 90% CI 2-sided [-1.67 to 0.98]
Statistical Analysis 4: Comparison: Latanoprost 0.005% and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 1 8 AM: Analysis was based on ANCOVA model for effect of taprenepag in combination with latanoprost compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.121, ANCOVA; LS mean difference = 1.26, 90% CI 2-sided [-0.07 to 2.59]
Statistical Analysis 5: Comparison: Latanoprost 0.005% and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; p = 0.039, ANCOVA; LS mean difference = 1.67, 90% CI 2-sided [0.34 to 2.99]
Statistical Analysis 6: Comparison: Latanoprost 0.005% and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; p = 0.220, ANCOVA; LS mean difference = 0.99, 90% CI 2-sided [-0.34 to 2.31]
Statistical Analysis 7: Comparison: Latanoprost Vehicle and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 7 8 AM: Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.098, ANCOVA; LS mean difference = 1.30, 90% CI 2-sided [0.01 to 2.59]
Statistical Analysis 8: Comparison: Latanoprost Vehicle and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.519, ANCOVA; LS mean difference = 0.50, 90% CI 2-sided [-0.77 to 1.77]
Statistical Analysis 9: Comparison: Latanoprost Vehicle and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.724, ANCOVA; LS mean difference = 0.27, 90% CI 2-sided [-1.00 to 1.55]
Statistical Analysis 10: Comparison: Latanoprost 0.005% and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 7 8 AM: Analysis was based on ANCOVA model for effect of taprenepag in combination with latanoprost compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.059, ANCOVA; LS mean difference = 1.46, 90% CI 2-sided [0.19 to 2.74]
Statistical Analysis 11: Comparison: Latanoprost 0.005% and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 2.71, 90% CI 2-sided [1.43 to 3.98]
Statistical Analysis 12: Comparison: Latanoprost 0.005% and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; p = 0.008, ANCOVA; LS mean difference = 2.09, 90% CI 2-sided [0.82 to 3.37]
Statistical Analysis 13: Comparison: Latanoprost Vehicle and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 7 10 AM: Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.068, ANCOVA; LS mean difference = 1.32, 90% CI 2-sided [0.13 to 2.51]
Statistical Analysis 14: Comparison: Latanoprost Vehicle and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.994, ANCOVA; LS mean difference = 0.01, 90% CI 2-sided [-1.16 to 1.18]
Statistical Analysis 15: Comparison: Latanoprost Vehicle and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.494, ANCOVA; LS mean difference = 0.50, 90% CI 2-sided [-0.70 to 1.69]
Statistical Analysis 16: Comparison: Latanoprost 0.005% and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 7 10 AM: Analysis was based on ANCOVA model for effect of taprenepag in combination with latanoprost compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.063, ANCOVA; LS mean difference = 1.39, 90% CI 2-sided [0.16 to 2.62]
Statistical Analysis 17: Comparison: Latanoprost 0.005% and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 16]; Test type: Superiority or Other; p = 0.004, ANCOVA; LS mean difference = 2.15, 90% CI 2-sided [0.95 to 3.34]
Statistical Analysis 18: Comparison: Latanoprost 0.005% and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 16]; Test type: Superiority or Other; p = 0.004, ANCOVA; LS mean difference = 2.17, 90% CI 2-sided [0.97 to 3.38]
Statistical Analysis 19: Comparison: Latanoprost Vehicle and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 7 1 PM: Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.038, ANCOVA; LS mean difference = 1.55, 90% CI 2-sided [0.32 to 2.77]
Statistical Analysis 20: Comparison: Latanoprost Vehicle and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 7 1 PM : Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.512, ANCOVA; LS mean difference = 0.48, 90% CI 2-sided [-0.72 to 1.68]
Statistical Analysis 21: Comparison: Latanoprost Vehicle and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p = 0.373, ANCOVA; LS mean difference = 0.66, 90% CI 2-sided [-0.56 to 1.89]
Statistical Analysis 22: Comparison: Latanoprost 0.005% and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 7 1 PM: Analysis was based on ANCOVA model for effect of taprenepag in combination with latanoprost compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.088, ANCOVA; LS mean difference = 1.31, 90% CI 2-sided [0.05 to 2.56]
Statistical Analysis 23: Comparison: Latanoprost 0.005% and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 22]; Test type: Superiority or Other; p = 0.004, ANCOVA; LS mean difference = 2.21, 90% CI 2-sided [0.98 to 3.44]
Statistical Analysis 24: Comparison: Latanoprost 0.005% and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 22]; Test type: Superiority or Other; p = 0.003, ANCOVA; LS mean difference = 2.33, 90% CI 2-sided [1.09 to 3.57]
Statistical Analysis 25: Comparison: Latanoprost Vehicle and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 7 4 PM: Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.010, ANCOVA; LS Mean Difference = 1.87, 90% CI 2-sided [0.69 to 3.04]
Statistical Analysis 26: Comparison: Latanoprost Vehicle and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p = 0.205, ANCOVA; LS mean difference = 0.89, 90% CI 2-sided [-0.27 to 2.05]
Statistical Analysis 27: Comparison: Latanoprost Vehicle and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p = 0.045, ANCOVA; LS mean difference = 1.44, 90% CI 2-sided [0.26 to 2.63]
Statistical Analysis 28: Comparison: Latanoprost 0.005% and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 7 4 PM: Analysis was based on ANCOVA model for effect of taprenepag in combination with latanoprost compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.005, ANCOVA; LS mean difference = 2.09, 90% CI 2-sided [0.88 to 3.31]
Statistical Analysis 29: Comparison: Latanoprost 0.005% and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 28]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 2.51, 90% CI 2-sided [1.33 to 3.70]
Statistical Analysis 30: Comparison: Latanoprost 0.005% and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 28]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS mean difference = 2.29, 90% CI 2-sided [1.10 to 3.48]
Statistical Analysis 31: Comparison: Latanoprost Vehicle and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 14 8 AM: Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.757, ANCOVA; LS mean difference = 0.27, 90% CI 2-sided [-1.15 to 1.69]
Statistical Analysis 32: Comparison: Latanoprost Vehicle and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p = 0.878, ANCOVA; LS mean difference = -0.13, 90% CI 2-sided [-1.54 to 1.27]
Statistical Analysis 33: Comparison: Latanoprost Vehicle and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; p = 0.780, ANCOVA; LS mean difference = -0.24, 90% CI 2-sided [-1.64 to 1.17]
Statistical Analysis 34: Comparison: Latanoprost 0.005% and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 14 8 AM: Analysis was based on ANCOVA model for effect of taprenepag in combination with latanoprost compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.670, ANCOVA; LS mean difference = 0.36, 90% CI 2-sided [-1.04 to 1.77]
Statistical Analysis 35: Comparison: Latanoprost 0.005% and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 34]; Test type: Superiority or Other; p = 0.021, ANCOVA; LS mean difference = 1.98, 90% CI 2-sided [0.58 to 3.38]
Statistical Analysis 36: Comparison: Latanoprost 0.005% and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 34]; Test type: Superiority or Other; p = 0.126, ANCOVA; LS mean difference = 1.31, 90% CI 2-sided [-0.10 to 2.71]
Statistical Analysis 37: Comparison: Latanoprost Vehicle and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 14 10 AM: Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.215, ANCOVA; LS mean difference = 0.97, 90% CI 2-sided [-0.32 to 2.26]
Statistical Analysis 38: Comparison: Latanoprost Vehicle and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p = 0.635, ANCOVA; LS mean difference = -0.37, 90% CI 2-sided [-1.65 to 0.91]
Statistical Analysis 39: Comparison: Latanoprost Vehicle and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; p = 0.934, ANCOVA; LS mean difference = -0.06, 90% CI 2-sided [-1.35 to 1.22]
Statistical Analysis 40: Comparison: Latanoprost 0.005% and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 14 10 AM: Analysis was based on ANCOVA model for effect of taprenepag in combination with latanoprost compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.478, ANCOVA; LS mean difference = 0.56, 90% CI 2-sided [-0.74 to 1.87]
Statistical Analysis 41: Comparison: Latanoprost 0.005% and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 40]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS mean difference = 2.57, 90% CI 2-sided [1.26 to 3.87]
Statistical Analysis 42: Comparison: Latanoprost 0.005% and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 40]; Test type: Superiority or Other; p = 0.013, ANCOVA; LS mean difference = 1.99, 90% CI 2-sided [0.68 to 3.30]
Statistical Analysis 43: Comparison: Latanoprost Vehicle and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 14 1 PM: Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.736, ANCOVA; LS mean difference = 0.27, 90% CI 2-sided [-1.04 to 1.57]
Statistical Analysis 44: Comparison: Latanoprost Vehicle and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p = 0.386, ANCOVA; LS mean difference = -0.68, 90% CI 2-sided [-1.96 to 0.61]
Statistical Analysis 45: Comparison: Latanoprost Vehicle and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 43]; Test type: Superiority or Other; p = 0.948, ANCOVA; LS mean difference = -0.05, 90% CI 2-sided [-1.35 to 1.24]
Statistical Analysis 46: Comparison: Latanoprost 0.005% and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 14 1 PM: Analysis was based on ANCOVA model for effect of taprenepag in combination with latanoprost compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.908, ANCOVA; LS mean difference = -0.09, 90% CI 2-sided [-1.41 to 1.22]
Statistical Analysis 47: Comparison: Latanoprost 0.005% and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 46]; Test type: Superiority or Other; p = 0.015, ANCOVA; LS mean difference = 1.97, 90% CI 2-sided [0.65 to 3.28]
Statistical Analysis 48: Comparison: Latanoprost 0.005% and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 46]; Test type: Superiority or Other; p = 0.046, ANCOVA; LS mean difference = 1.60, 90% CI 2-sided [0.29 to 2.92]
Statistical Analysis 49: Comparison: Latanoprost Vehicle and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 14 4 PM: Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.042, ANCOVA; LS mean difference = 1.60, 90% CI 2-sided [0.31 to 2.89]
Statistical Analysis 50: Comparison: Latanoprost Vehicle and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p = 0.940, ANCOVA; LS mean difference = 0.06, 90% CI 2-sided [-1.22 to 1.34]
Statistical Analysis 51: Comparison: Latanoprost Vehicle and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 49]; Test type: Superiority or Other; p = 0.114, ANCOVA; LS mean difference = 1.24, 90% CI 2-sided [-0.05 to 2.53]
Statistical Analysis 52: Comparison: Latanoprost 0.005% and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 14 4 PM: Analysis was based on ANCOVA model for effect of taprenepag in combination with latanoprost compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.228, ANCOVA; LS mean difference = 0.97, 90% CI 2-sided [-0.35 to 2.28]
Statistical Analysis 53: Comparison: Latanoprost 0.005% and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 52]; Test type: Superiority or Other; p = 0.005, ANCOVA; LS mean difference = 2.29, 90% CI 2-sided [0.98 to 3.60]
Statistical Analysis 54: Comparison: Latanoprost 0.005% and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 52]; Test type: Superiority or Other; p = 0.063, ANCOVA; LS mean difference = 1.48, 90% CI 2-sided [0.17 to 2.79]
Statistical Analysis 55: Comparison: Latanoprost Vehicle and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 28 8 AM: Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.562, ANCOVA; LS mean difference = 0.50, 90% CI 2-sided [-0.92 to 1.91]
Statistical Analysis 56: Comparison: Latanoprost Vehicle and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p = 0.431, ANCOVA; LS mean difference = 0.67, 90% CI 2-sided [-0.73 to 2.07]
Statistical Analysis 57: Comparison: Latanoprost Vehicle and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 55]; Test type: Superiority or Other; p = 0.795, ANCOVA; LS mean difference = 0.22, 90% CI 2-sided [-1.18 to 1.62]
Statistical Analysis 58: Comparison: Latanoprost 0.005% and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 28 8 AM: Analysis was based on ANCOVA model for effect of taprenepag in combination with latanoprost compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.032, ANCOVA; LS mean difference = 1.83, 90% CI 2-sided [0.43 to 3.23]
Statistical Analysis 59: Comparison: Latanoprost 0.005% and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 58]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS mean difference = 2.73, 90% CI 2-sided [1.34 to 4.13]
Statistical Analysis 60: Comparison: Latanoprost 0.005% and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 58]; Test type: Superiority or Other; p = 0.017, ANCOVA; LS mean difference = 2.04, 90% CI 2-sided [0.64 to 3.44]
Statistical Analysis 61: Comparison: Latanoprost Vehicle and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 28 10 AM: Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.124, ANCOVA; LS mean difference = 1.26, 90% CI 2-sided [-0.09 to 2.60]
Statistical Analysis 62: Comparison: Latanoprost Vehicle and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p = 0.920, ANCOVA; LS mean difference = 0.08, 90% CI 2-sided [-1.25 to 1.41]
Statistical Analysis 63: Comparison: Latanoprost Vehicle and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 61]; Test type: Superiority or Other; p = 0.887, ANCOVA; LS mean difference = -0.12, 90% CI 2-sided [-1.46 to 1.22]
Statistical Analysis 64: Comparison: Latanoprost 0.005% and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 28 10 AM: Analysis was based on ANCOVA model for effect of taprenepag in combination with latanoprost compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.083, ANCOVA; LS mean difference = 1.42, 90% CI 2-sided [0.08 to 2.77]
Statistical Analysis 65: Comparison: Latanoprost 0.005% and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 64]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS mean difference = 2.65, 90% CI 2-sided [1.29 to 4.01]
Statistical Analysis 66: Comparison: Latanoprost 0.005% and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 64]; Test type: Superiority or Other; p = 0.006, ANCOVA; LS mean difference = 2.30, 90% CI 2-sided [0.94 to 3.66]
Statistical Analysis 67: Comparison: Latanoprost Vehicle and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 28 1 PM: Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.533, ANCOVA; LS mean difference = 0.49, 90% CI 2-sided [-0.80 to 1.78]
Statistical Analysis 68: Comparison: Latanoprost Vehicle and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.985, ANCOVA; LS mean difference = -0.02, 90% CI 2-sided [-1.29 to 1.26]
Statistical Analysis 69: Comparison: Latanoprost Vehicle and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 67]; Test type: Superiority or Other; p = 0.665, ANCOVA; LS mean difference = 0.34, 90% CI 2-sided [-0.95 to 1.62]
Statistical Analysis 70: Comparison: Latanoprost 0.005% and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 28 1 PM: Analysis was based on ANCOVA model for effect of taprenepag in combination with latanoprost compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.276, ANCOVA; LS mean difference = 0.86, 90% CI 2-sided [-0.44 to 2.15]
Statistical Analysis 71: Comparison: Latanoprost 0.005% and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 70]; Test type: Superiority or Other; p = 0.004, ANCOVA; LS mean difference = 2.34, 90% CI 2-sided [1.04 to 3.65]
Statistical Analysis 72: Comparison: Latanoprost 0.005% and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 70]; Test type: Superiority or Other; p = 0.011, ANCOVA; LS mean difference = 2.04, 90% CI 2-sided [0.74 to 3.35]
Statistical Analysis 73: Comparison: Latanoprost Vehicle and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 28 4 PM: Analysis was based on ANCOVA model for effect of taprenepag alone compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.033, ANCOVA; LS mean difference = 1.78, 90% CI 2-sided [0.41 to 3.14]
Statistical Analysis 74: Comparison: Latanoprost Vehicle and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.302, ANCOVA; LS mean difference = 0.84, 90% CI 2-sided [-0.50 to 2.19]
Statistical Analysis 75: Comparison: Latanoprost Vehicle and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 73]; Test type: Superiority or Other; p = 0.255, ANCOVA; LS mean difference = 0.94, 90% CI 2-sided [-0.42 to 2.30]
Statistical Analysis 76: Comparison: Latanoprost 0.005% and Taprenepag 0.005% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); Change at Day 28 4 PM: Analysis was based on ANCOVA model for effect of taprenepag in combination with latanoprost compared to latanoprost alone on IOP reduction from baseline with treatment and baseline IOP as covariates; Test type: Superiority or Other; p = 0.198, ANCOVA; LS mean difference = 1.08, 90% CI 2-sided [-0.30 to 2.46]
Statistical Analysis 77: Comparison: Latanoprost 0.005% and Taprenepag 0.01% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 76]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS mean difference = 2.68, 90% CI 2-sided [1.30 to 4.06]
Statistical Analysis 78: Comparison: Latanoprost 0.005% and Taprenepag 0.015% (Stage II) vs Latanoprost 0.005% and Taprenepag Vehicle (Stage II); [analysis description as in outcome 8, analysis 76]; Test type: Superiority or Other; p = 0.046, ANCOVA; LS mean difference = 1.68, 90% CI 2-sided [0.30 to 3.06]

9. Secondary Outcome: Percentage of Participants Reaching and Maintaining Target Intra Ocular Pressure (IOP): Stage I
Description: Percentage of participants who reached an IOP of less than or equal to (<=) 18 mmHg by post-eligibility visit (Day 1) and maintained an IOP <= 18 mm Hg across all post-eligibility visits in Stage I were reported. IOP was measured using Goldmann applanation tonometer.
Time Frame: Stage I: Day 1 up to Day 14
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Taprenepag 0.0025% (Stage I) | Taprenepag 0.005% (Stage I) | Taprenepag 0.01% (Stage I) | Taprenepag 0.015% (Stage I) | Taprenepag 0.02% (Stage I) | Taprenepag 0.03% (Stage I) | Taprenepag Vehicle (Stage I)
Number analyzed (Participants) | 9 | 9 | 9 | 10 | 9 | 9 | 12
percentage of participants | 0.0 | 11.1 | 11.1 | 0.0 | 11.1 | 22.2 | 0.0

10. Secondary Outcome: Percentage of Participants Reaching and Maintaining Target Intra Ocular Pressure (IOP): Stage II
Description: Percentage of participants who reached an IOP <= 18 mmHg by post-eligibility visit (Day 1) and maintained an IOP <= 18 mm Hg across all post-eligibility visits in Stage II were reported. IOP was measured using Goldmann applanation tonometer.
Time Frame: Stage II: Day 1 up to Day 28
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Latanoprost Vehicle and Taprenepag 0.005% (Stage II) | Latanoprost Vehicle and Taprenepag 0.01% (Stage II) | Latanoprost Vehicle and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag 0.005% (Stage II) | Latanoprost 0.005% and Taprenepag 0.01% (Stage II) | Latanoprost 0.005% and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag Vehicle (Stage II)
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 36 | 36 | 35
percentage of participants | 22.9 | 2.8 | 13.9 | 8.3 | 38.9 | 16.7 | 5.7

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Taprenepag 0.0025% (Stage I) | Taprenepag 0.005% (Stage I) | Taprenepag 0.01% (Stage I) | Taprenepag 0.015% (Stage I) | Taprenepag 0.02% (Stage I) | Taprenepag 0.03% (Stage I) | Taprenepag Vehicle (Stage I) | Latanoprost Vehicle and Taprenepag 0.005% (Stage II) | Latanoprost Vehicle and Taprenepag 0.01% (Stage II) | Latanoprost Vehicle and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag 0.005% (Stage II) | Latanoprost 0.005% and Taprenepag 0.01% (Stage II) | Latanoprost 0.005% and Taprenepag 0.015% (Stage II) | Latanoprost 0.005% and Taprenepag Vehicle (Stage II)
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/10 | 0/9 | 0/9 | 0/12 | 0/35 | 1/36 | 2/36 | 0/36 | 0/36 | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 3/9 | 3/9 | 0/9 | 5/10 | 5/9 | 9/9 | 4/12 | 18/35 | 20/36 | 27/36 | 24/36 | 27/36 | 26/36 | 15/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Taprenepag 0.0025% (Stage I) (N=9) | Taprenepag 0.005% (Stage I) (N=9) | Taprenepag 0.01% (Stage I) (N=9) | Taprenepag 0.015% (Stage I) (N=10) | Taprenepag 0.02% (Stage I) (N=9) | Taprenepag 0.03% (Stage I) (N=9) | Taprenepag Vehicle (Stage I) (N=12) | Latanoprost Vehicle and Taprenepag 0.005% (Stage II) (N=35) | Latanoprost Vehicle and Taprenepag 0.01% (Stage II) (N=36) | Latanoprost Vehicle and Taprenepag 0.015% (Stage II) (N=36) | Latanoprost 0.005% and Taprenepag 0.005% (Stage II) (N=36) | Latanoprost 0.005% and Taprenepag 0.01% (Stage II) (N=36) | Latanoprost 0.005% and Taprenepag 0.015% (Stage II) (N=36) | Latanoprost 0.005% and Taprenepag Vehicle (Stage II) (N=35)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Taprenepag 0.0025% (Stage I) (N=9) | Taprenepag 0.005% (Stage I) (N=9) | Taprenepag 0.01% (Stage I) (N=9) | Taprenepag 0.015% (Stage I) (N=10) | Taprenepag 0.02% (Stage I) (N=9) | Taprenepag 0.03% (Stage I) (N=9) | Taprenepag Vehicle (Stage I) (N=12) | Latanoprost Vehicle and Taprenepag 0.005% (Stage II) (N=35) | Latanoprost Vehicle and Taprenepag 0.01% (Stage II) (N=36) | Latanoprost Vehicle and Taprenepag 0.015% (Stage II) (N=36) | Latanoprost 0.005% and Taprenepag 0.005% (Stage II) (N=36) | Latanoprost 0.005% and Taprenepag 0.01% (Stage II) (N=36) | Latanoprost 0.005% and Taprenepag 0.015% (Stage II) (N=36) | Latanoprost 0.005% and Taprenepag Vehicle (Stage II) (N=35)
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abnormal sensation in eye, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal sensation in eye, RIGHT EYE, STUDY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenopia, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract nuclear, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chalazion, LEFT EYE, STUDY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chorioretinopathy, RIGHT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctival haemorrhage, LEFT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage, RIGHT EYE, STUDY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctival hyperaemia, BOTH EYES (Eye disorders) | 1 | 2 | 0 | 1 | 0 | 5 | 3 | 10 | 10 | 11 | 13 | 13 | 13 | 9
Conjunctival hyperaemia, LEFT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Conjunctival hyperaemia, LEFT EYE, STUDY EYE (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Conjunctival hyperaemia, RIGHT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Conjunctival hyperaemia, RIGHT EYE, STUDY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Corneal disorder, BOTH EYES (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0
Corneal erosion, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1
Corneal erosion, LEFT EYE, STUDY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Corneal erosion, RIGHT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Corneal oedema, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Dry eye, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Erythema of eyelid, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Extraocular muscle disorder, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye discharge, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye inflammation, LEFT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 3 | 5 | 3 | 5
Eye pain, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 3 | 3 | 3 | 6 | 1
Eye pain, LEFT EYE, STUDY EYE (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain, RIGHT EYE, STUDY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pruritus, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 3 | 2 | 2 | 1
Eyelid oedema, LEFT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eyelids pruritus, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foreign body sensation in eyes, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foreign body sensation in eyes, LEFT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foreign body sensation in eyes, RIGHT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypermetropia, LEFT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Iritis, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 3 | 1 | 1 | 4 | 0
Iritis, LEFT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Iritis, LEFT EYE, STUDY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Iritis, RIGHT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Iritis, RIGHT EYE, STUDY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Lacrimation increased, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Macular oedema, LEFT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myodesopsia, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myopia, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ocular discomfort, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Ocular hyperaemia, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Ocular hyperaemia, LEFT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia, RIGHT EYE, STUDY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Open angle glaucoma, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photophobia, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 1 | 3 | 4 | 0 | 5 | 5 | 12 | 7 | 7 | 15 | 1
Photophobia, LEFT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 3 | 4 | 5 | 1 | 3 | 0
Vision blurred, LEFT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred, RIGHT EYE, STUDY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual acuity reduced, BOTH EYES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Visual acuity reduced, LEFT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Visual acuity reduced, LEFT EYE, STUDY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual acuity reduced, RIGHT EYE, FELLOW EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Instillation site irritation, BOTH EYES (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1
Instillation site pain, BOTH EYES (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sensation of foreign body, BOTH EYES (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis viral, RIGHT EYE, FELLOW EYE (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Corneal staining, BOTH EYES (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Corneal staining, LEFT EYE, FELLOW EYE (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Corneal staining, RIGHT EYE, STUDY EYE (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Headache, BOTH EYES (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Migraine, BOTH EYES (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual field defect, BOTH EYES (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.